CLINICAL TRIAL: NCT06987786
Title: Differences in Mechanistic Measures (Oxytocin and Cortisol) of Therapeutic Alliance Between A Talk-Based Therapy and Soft-Tissue Mobilization in Individuals With Chronic Spinal Pain
Acronym: COTHA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Pro00118076
Record Dates: First submitted 2025-05-06; First posted 2025-05-23 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-05

CONDITIONS: Spine; Low Back Pain; Neck Pain
Keywords: Oxytocin; Cortisol; spinal pain
MeSH Terms: conditions — Low Back Pain; Neck Pain | interventions — Massage

STUDY DESIGN:
Intervention Model Description: This proposal involves a randomized, cross-over mechanistic clinical trial that includes a cohort of participants with chronic spine pain. A randomized, cross-over mechanistic trial is useful because it allows each participant to serve as their own control, reducing variability and increasing the statistical power to detect treatment effects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage, then talk-based therapy (Experimental): Subjects will be randomized to receive massage for one session, then will receive talk-based therapy after a two week washout period.
  Interventions: Other: Massage; Other: Talk-based therapy
- Talk-based therapy, then massage (Experimental): Subjects will be randomized to receive talk-based therapy first, then after a 2 week wash out period will receive a massage threatment
  Interventions: Other: Massage; Other: Talk-based therapy

INTERVENTIONS:
Other: Massage — Soft tissue mobilization (STM), also known as massage, is a form of manual therapy. STM consists of many different categories of treatment, but all involve a "hand's on" application. During the session, the Dr. Cook will use techniques such as kneading, stretching, and deep tissue manipulation to target the affected areas. The total time of application will be 30 minutes. This "hands-on" approach is theorized to reduce muscle tension, improve blood circulation, and promote relaxation. STM stimulates the release of endorphins and serotonin, which are natural painkillers and mood enhancers.
Other: Talk-based therapy — Talk based therapy includes an innovative, evidence-based psychosocial therapy designed to provide rapid and effective pain management for individuals suffering from chronic pain. This single-session, intervention equips patients with essential pain relief skills through a combination of cognitive behavioral therapy (CBT) techniques, mindfulness principles, and pain neuroscience education. The program focuses on teaching patients how to identify and reframe distressing thoughts, practice relaxation techniques, and develop personalized pain management plans.

SUMMARY:
The goal of this randomized cross-over mechanistic trial is to compare pre- and post-level cortisol and oxytocin changes in patients with chronic spine pain who receive either a hand's on (massage) or a hand's off (talk-based) approach. The study plans to address two primary aims.

Specific Aim One: Directly compare pre- and post-session oxytocin and cortisol levels across two sessions of massage and talk-based therapy. Hypothesis 1: It is expected that in both treatments, oxytocin will increase and cortisol will decrease, demonstrating no significant between-group differences in hormone levels.

Specific Aim Two: The study plans to compare pre- and post-session oxytocin and cortisol change scores a therapeutic alliance (TA) scale change scores and PROMIS patient-reported outcomes associated with pain, depression, and disability. Hypothesis 2a: It is projected that there will be moderate +/- relationships (R>.4) between the therapeutic alliance change score and oxytocin and cortisol levels, suggesting that the hormones moderately reflect the construct associated with TA. Hypothesis 2b: It is expected that there will be weak (R>.1) +/-relationships between hormone measures and PROMIS pain/disability/depression measures, which reflects similar findings to preliminary work.

Participants will participant in a massage based treatment and a talk-based treatment approach. Participants will also complete patient report outcomes and will receive a total of four salivary swabs.

DETAILED DESCRIPTION:
Recruitment at Duke University: Recruitment will follow a well-versed, successful process at Duke University. MaestroCare will be used to identify, recruit, and conduct this research study. Participants will be invited to participate in this study via a MyChart patient portal invitation sent by a clinical research coordinator (CRC). The CRC will screen participants for eligibility via telephone encounter. Prior to obtaining consent, participants will be screened for medical conditions that may influence hormone levels during the study (e.g., Cushing's Syndrome, Addison's Disease, etc.), use of medications (e.g., steroids, antidepressants, or hormonal treatments) that could influence the results, and exclude participants if necessary, and previously diagnosed conditions or factors known to affect cortisol or oxytocin levels, such as chronic stress disorders, hormonal imbalances, or pregnancy. After obtaining consent and prior to treatment, the study will screen for potential STM contraindications or other clinical safety considerations (i.e., infection, skin lesions, etc) using a limited systems-screening to rule out pertinent clinical contraindications to STM (e.g., radiculopathy, fracture, etc.).

Participants: Individuals with CSP (3 months or greater), who are 18 years of age and older and who experience persistent pain of ≥3 on a 10-point scale for the majority of days during the previous 3-months will be eligible for the study. The study operationally defines chronic pain using the International Association of the Study of Pain (IASP) pragmatic criteria of pain lasting for 3 months or more that cannot be attributed to another diagnosis or condition.

Variables: In addition to pertinent demographics and patient characteristics, the study will capture baseline PROMIS pain interference, pain intensity, depression, and physical function values. Onsite, to improve the likelihood that hormone related changes are not influenced by external factors, the study will capture a Perceived Stress Scale (PSS), which measures subjective stress levels, State-Trait Anxiety Inventory (STAI), which assesses temporary and long-term anxiety states, blood pressure and pulse prior to each visit. For the PSS, a score of 27 or above is typically considered high. For the STAI, a score above 60 is often considered high, signaling significant anxiety. If individuals score high in either measure, the participants will be rescheduled. Those with Blood pressure: ≥140/90 mmHg and a heart rate >100bpm will be asked to reschedule.

The study's primary variables of interest in the study involve cortisol and oxytocin levels. The study will capture 525 μL salivary concentrations of oxytocin and cortisol through a SalivaBio Oral Swab (SOS) Method. Testing will be completed with Salimetrics Assay Kits. The study will also capture the self-report WAI short-form and the PROMIS pain interference, pain intensity, and physical function measures at baseline and after completion of both visits.

Interventions: After describing the study design and purpose, participants will be randomized into a single treatment of STM-first or a single treatment of ER-first. All treatments will be provided by Dr. Cook, a licensed physical therapist with 35 years of clinical experience and fellowship-level training in STM (e.g., manual therapies) and a 2.5-year post-professional, certification-level training in chronic pain management/psychologically informed practice. A designated clinical research coordinator (CRC) and Dr. Cook will be responsible for screening of each applicant to ensure the participants are appropriate and safe for study inclusion.

ELIGIBILITY:
Inclusion Criteria include:

* Individuals with chronic spine pain (3 months or greater) (and);
* who are 18 years of age and older (and)
* who experience persistent pain of ≥3 on a 10-point scale for the majority of days during the previous 3-months

(The study operationally defines chronic pain using the International Association of the Study of Pain (IASP) pragmatic criteria of pain lasting for 3 months or more that cannot be attributed to another diagnosis or condition).

-

Exclusion Criteria include:

* Participants with medical conditions that may influence hormone levels during the study (e.g., Cushing's Syndrome, Addison's Disease, etc.) (or),
* Use of medications (e.g., steroids, antidepressants, or hormonal treatments) that could influence the results (or)
* Previously diagnosed conditions or factors known to affect cortisol or oxytocin levels, such as chronic stress disorders, hormonal imbalances, or pregnancy.

(After obtaining consent and prior to treatment), the study will screen for potential massage contraindications or other clinical safety considerations and will exclude if:

* participants have infection, skin lesions, (or)
* Fractures in the region of the massage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Cortisol changes | Day 1 and day 15
  The study will capture 525 μL salivary concentrations cortisol through a SalivaBio Oral Swab (SOS) Method. Testing will be completed with Salimetrics Assay Kits.
Oxytocin changes | Day 1 and day 15
  The study will capture 525 μL salivary concentrations of oxytocin through a SalivaBio Oral Swab (SOS) Method. Testing will be completed with Salimetrics Assay Kits.

SECONDARY OUTCOMES:
Therapeutic alliance | Day 1 and day 15
  Working Alliance Inventory (WAI) short-form. The Working Alliance Inventory (WAI) measures three important aspects of the therapeutic alliance: 1. Agreement about the therapeutic tasks, 2. Agreement about the therapeutic goals, and 3. The affective bond between clinician and client. The WAI short-form is scored by adding up individual item responses, which are rated on a 5-point Likert scale (1=rarely or never to 5=always). The Working Alliance Inventory-Short (WAI-S) has a total score ranging from 12 to 84. A higher score indicates a stronger working alliance between a patient and therapist.
PROMIS pain interference | Day 1 and day 15
  The PROMIS Pain Interference (PROMIS-PI) measure assesses the extent to which pain affects a person's daily life, specifically their ability to engage in social, cognitive, emotional, physical, and recreational activities. It's a widely used instrument within the PROMIS (Patient-Reported Outcomes Measurement Information System) initiative, a set of tools for measuring patient-reported outcomes in various health conditions. The PROMIS Pain Interference (PI) scale, particularly the 4-item short form (4a), measures how much pain interferes with an individual's activities over the past 7 days. Each question is answered on a 5-point scale (1=never to 5=almost always), and the total score is calculated by summing the individual item scores. For the 4-item short form, the total raw score range is 4 to 20, with higher scores indicating greater pain interference. PROMIS also uses a T-score metric, where the mean is 50 and the standard deviation is 10.
PROMIS Pain intensity | Day 1 and day 15
  The PROMIS Pain Intensity measure assesses how much pain a person is experiencing. It uses a numeric rating scale (NRS) where individuals rate their pain on a scale from 0 (no pain) to 10 (worst possible pain). The PROMIS Pain Intensity measure is part of the broader Patient-Reported Outcomes Measurement Information System (PROMIS) initiative, which aims to develop standardized, reliable, and valid tools for measuring patient-reported outcomes.
PROMIS Depression | Day 1 and day 15
  The PROMIS Depression measure is a tool used to assess depression, specifically focusing on affective and cognitive symptoms like sadness, guilt, and self-criticism. It's part of the Patient-Reported Outcomes Measurement Information System (PROMIS), a collection of measures designed to evaluate patient-reported outcomes. PROMIS Depression 4 scale measures depression severity using a four-item questionnaire. Each item is rated on a scale, and the total score is the sum of these ratings, ranging from 4 to 20. Higher scores indicate more severe depression. It's important to note that PROMIS scales, including the 4-item depression scale, also use a T-score system, which is a standardized score with a mean of 50 and a standard deviation of 10.
PROMIS physical function | Day 1 and day 15
  The PROMIS Physical Function 4 scale is measured using a series of questions assessing a person's ability to perform various physical tasks, with responses scored on a 5-point Likert scale. The raw score from these responses is then converted to a standardized T-score on a scale of 0 to 100, with a mean of 50 and a standard deviation of 10. The total score is the final T-score.

CONTACTS AND LOCATIONS:
Overall Officials: Chad E Cook, Principal Investigator — Duke University
Locations (1):
- CORE 2200 West Main Street, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No